## STUDY PROTOCOL

THE IMPACT OF LOCAL VS. SYSTEMIC ADJUVANT ANTIBIOTICS DURING NON-SURGICAL PERIODONTITIS THERAPY ON CLINICAL PARAMETERS, BACTERIAL COUNT AND CYTOKINE LEVELS – A RANDOMIZED CLINICAL TRIAL

NCT05608564

Date: 15.1.2022.

#### **Background and objectives**

Periodontitis is a chronic inflammatory disease that leads to progressive destruction of periodontal tissues and tooth-supporting structures, primarily driven by microbial dysbiosis and an altered host immune response (1,2). The excessive accumulation of immunomodulatory cells due to inadequate immune regulation contributes to alveolar bone loss (3). Among key inflammatory mediators, tumor necrosis factor-alpha (TNF- $\alpha$ ) plays a crucial role in initiating immune responses against periodontal pathogens and promoting bone resorption (4-6). Similarly, interleukin-17 (IL-17) has been linked to both immune defense and pathological bone loss through neutrophil recruitment and activation of osteoclasts (7,8).

Non-surgical periodontal therapy (NSPT) is the first-line treatment aimed at reducing bacterial burden and controlling inflammation through mechanical debridement (9). Although effective, NSPT alone may not be sufficient for optimal outcomes, leading to the adjunctive use of systemic antibiotics, particularly amoxicillin, and metronidazole, which have demonstrated significant clinical benefits in younger individuals with generalized stage III periodontitis (10-12). The combination of these antibiotics has been associated with favorable shifts in the subgingival microbiome and long-term clinical improvements (13). However, while in vitro studies suggest metronidazole can inhibit TNF- $\alpha$  production, clinical evidence remains inconsistent (14,15). Additionally, local antibiotic delivery has shown mixed results, with some studies reporting clinical benefits while others limit its use to maintenance therapy or persistent deep pockets (16-18).

Given the conflicting evidence, the primary objective of this study is to compare the clinical outcomes of systemic versus locally delivered adjuvant antibiotics during NSPT at baseline and after six months. The secondary objective is to evaluate their effects on total bacterial load and the relative expression levels of key pro-inflammatory mediators such as TNF- $\alpha$  and IL-17.

#### Material and methods

#### Study design and participants

This randomized clinical study will include 38 patients diagnosed with periodontitis stage III. The investigation will be conducted at the Department of Periodontology and Oral Medicine, at the School of Dental Medicine, University of Belgrade. The laboratory part of the research will be carried out at the Department of Human Genetics, at the School of Dental Medicine, University of Belgrade. This research initiation is approved by the Ethical Committee of the School of Dental Medicine, University of Belgrade (No 36/6). Patients will be divided into two groups. The test group will consist of 19 patients who will receive a local antibiotic (LA group), while the control group will consist of 19 patients who will be prescribed systemic antibiotic therapy (SA group). The division of patients into groups will be done using randomization envelopes after the diagnostic procedure.

Participants will be eligible for inclusion if they meet the following inclusion criteria:

- Individuals aged 18–40 years
- Willingness to participate in the research, comply with all study protocols, and provide signed informed consent
- Diagnosis of active periodontitis stage III according to the latest classification (1)
- Non-smokers or light smokers (≤10 cigarettes/day)

#### Exclusion Criteria:

- Presence of systemic diseases affecting periodontal or bone metabolism (e.g., uncontrolled diabetes, cancer, immunodeficiency, metabolic bone diseases)
- Ongoing treatment with immunosuppressive, anti-resorptive, or anti-inflammatory medications
- Known penicillin allergy
- History of periodontal therapy within the last six months
- Use of local or systemic antimicrobials in the past six months
- Use of oral anti-plaque mouthwash within one month before the study
- Alcohol or drug abuse
- · Pregnancy or lactation

# Data collection and sampling

Upon clinical examination, clinical periodontal parameters such as pocket probing depth (PPD), clinical attachment level (CAL), bleeding on probing (BOP), and plaque index (PI) will be recorded for each patient around every tooth. Prior to treatment, subgingival crevicular fluid will be sampled with paper points from periodontal pockets for laboratory analysis.

Sampling will be performed as follows: first, a relatively dry working field will be established using paper water rollers and air jets. Then, three paper points (number 30 – marked in blue) will be applied for 30 seconds in the periodontal pocket area of the selected premolar/molar tooth with a depth of more than 5 mm. The procedure will be repeated immediately in the same region to obtain duplicate samples. After that, the paper points will be placed in Eppendorf tubes and immediately transported to the basic research laboratory, where they will be stored at a temperature of –80 degrees Celsius for subsequent microbiological and molecular analyses.

### Non-surgical periodontal therapy and antibiotic administration

After sampling, all patients will undergo a non-surgical phase of periodontal therapy (NSPT) following a Full-Mouth Disinfection protocol (19). Six months after the NSPT, at follow-up, the detection of clinical parameters and the sampling procedure will be repeated.

In the LA group, a combination of piperacillin and tazobactam in gel form (Gelcide ®, Italmed MedTechDental, Florence, Italy) designed for subgingival use will be applied locally. The local antibiotic will be administered into the periodontal pockets using a syringe and a flexible blunt needle, 24 hours after NSPT. The administration will be done by quadrants, following the principles of a dry work field, and after application, the dry field will be maintained for five minutes. After this procedure, the patient will be instructed not to rinse the oral cavity for 15 minutes.

For systemic use in the SA group, patients will receive a combination of Amoxicillin (Amoxicillin  $^{\circ}$ , 500 mg, three times a day, for seven days) and Metronidazole (Orvagyl  $^{\circ}$ , 400 mg, three times a day, for seven days) for oral use after NSPT is completed (11).

#### **Laboratory Analyses**

Total bacterial count (TBC) and relative expression levels (REL) of proinflammatory cytokines TNF-  $\alpha$  and IL-17 will be detected using quantitative real-time polymerase chain reaction (qPCR) in a basic research laboratory at the Department of Human Genetics, at the School of Dental Medicine, University of Belgrade (20, 21).

#### **Laboratory analyses**

Total bacterial count (TBC) and relative expression levels (REL) of proinflammatory cytokines TNF-  $\alpha$  and IL-17 will be detected using quantitative real-time polymerase chain reaction (qPCR) in a basic research laboratory at the Department of Human Genetics, at the School of Dental Medicine, University of Belgrade (20, 21).

### Statistical analyses

All statistical analyses will be performed on an intention-to-treat basis, with no expected dropouts during the observational period. Data analysis will be conducted using GraphPad Prism 9.0 (GraphPad, San Diego, CA, USA) and Statistical Package for Social Science (SPSS, version 26.0; SPSS Inc., Chicago, IL, USA). For numerical data, mean values, medians, standard deviations (SD), and ranges will be used for descriptive statistics.

The Kolmogorov–Smirnov normality test will be applied to examine the distribution of outcome variables. Depending on the distribution, paired Student's t-test or Wilcoxon signed-rank test will be used to compare baseline and six-month follow-up measurements between treatment groups. Repeated measures ANOVA with Bonferroni correction or Friedman and Wilcoxon signed-rank test will be used for within-group comparisons. Statistical significance will be set at p < 0.05.

#### References

- 1. Papapanou PN, Sanz M, Buduneli N, et al. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. Jun 2018;89:S173-S182. doi:10.1002/jper.17-0721
- 2. Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Clin Periodontol. Jun 2018;45:S149-S161. doi:10.1111/jcpe.12945
- 3. Tompkins KA. The osteoimmunology of alveolar bone loss. Connect Tissue Res. Mar 2016;57(2):69-90. doi:10.3109/03008207.2016.1140152
- 4. de Oliveira RR, Schwartz-Filho HO, Novaes AB, et al. Antimicrobial photodynamic therapy in the non-surgical treatment of aggressive periodontitis: cytokine profile in gingival crevicular fluid, preliminary results. J Periodontol. Jan 2009;80(1):98-105. doi:10.1902/jop.2009.070465
- 5. Gomes FI, Aragão MG, Barbosa FC, Bezerra MM, de Paulo Teixeira Pinto V, Chaves HV. Inflammatory Cytokines Interleukin- $1\beta$  and Tumour Necrosis Factor- $\alpha$  Novel Biomarkers for the Detection of Periodontal Diseases: a Literature Review. J Oral Maxillofac Res. Apr-Jun 2016;7(2):e2. doi:10.5037/jomr.2016.7202
- 6. Zhao BH. TNF and Bone Remodeling. Curr Osteoporos Rep. Jun 2017;15(3):126-134. doi:10.1007/s11914-017-0358-z
- 7. Abusleme L, Moutsopoulos NM. IL-17: overview and role in oral immunity and microbiome. Oral Diseases. Oct 2017;23(7):854-865. doi:10.1111/odi.12598
- 8. Moutsopoulos NM, Lionakis MS, Hajishengallis G. Inborn errors in immunity: unique natural models to dissect oral immunity. J Dent Res. Jun 2015;94(6):753-8. doi:10.1177/0022034515583533
- 9. Suvan J, Leira Y, Moreno Sancho FM, Graziani F, Derks J, Tomasi C. Subgingival instrumentation for treatment of periodontitis. A systematic review. J Clin Periodontol. Jul 2020;47 Suppl 22:155-175. doi:10.1111/jcpe.13245
- 10. Teughels W, Feres M, Oud V, Martín C, Matesanz P, Herrera D. Adjunctive effect of systemic antimicrobials in periodontitis therapy: A systematic review and meta-analysis. J Clin Periodontol. Jul 2020;47 Suppl 22:257-281. doi:10.1111/jcpe.13264
- 11. Sanz M, Herrera D, Kebschull M, et al. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. Jul 2020;47 Suppl 22(Suppl 22):4-60. doi:10.1111/jcpe.13290
- 12. Eickholz P, Koch R, Göde M, et al. Clinical benefits of systemic amoxicillin/metronidazole may depend on periodontitis stage and grade: An exploratory sub-analysis of the ABPARO trial. J Clin Periodontol. Sep 2023;50(9):1239-1252. doi:10.1111/jcpe.13838
- 13. Feres M, Figueiredo LC, Soares GMS, Faveri M. Systemic antibiotics in the treatment of periodontitis. Periodontol 2000. 2015;67(1):131-186.
- 14. Rizzo A, Paolillo R, Guida L, Annunziata M, Bevilacqua N, Tufano MA. Effect of metronidazole and modulation of cytokine production on human periodontal ligament cells. Int Immunopharmacol. Jul 2010;10(7):744-50. doi:10.1016/j.intimp.2010.04.004
- 15. Aral K, Aral CA, Kapila Y. Six-month clinical outcomes of non-surgical periodontal treatment with antibiotics on apoptosis markers in aggressive periodontitis. Oral Dis. Apr 2019;25(3):839-847. doi:10.1111/odi.13032

- 16. Herrera D, Matesanz P, Martín C, Oud V, Feres M, Teughels W. Adjunctive effect of locally delivered antimicrobials in periodontitis therapy: A systematic review and meta-analysis. J Clin Periodontol. 2020;47:239-256. doi: 10.1111/jcpe.13230
- 17. Rovai ES, Souto ML, Ganhito JA, Holzhausen M, Chambrone L, Pannuti CM. Efficacy of Local Antimicrobials in the Non-Surgical Treatment of Patients With Periodontitis and Diabetes: A Systematic Review. J Periodontol. Dec 2016;87(12):1406-1417. doi:10.1902/jop.2016.160214
- 18. Hussein I, Ranka M, Gilbert A, Davey K. Locally delivered antimicrobials in the management of periodontitis: a critical review of the evidence for their use in practice. Dent Update. Oct 2007;34(8):494-6, 499-502, 505-6. doi:10.12968/denu.2007.34.8.494
- 19. Heitz-Mayfield LJA, Lang NP. Surgical and nonsurgical periodontal therapy. Learned and unlearned concepts. Periodontol 2000. Jun 2013;62:218-231. doi:10.1111/prd.12008
- 20. Brajović G, Popović B, Puletić M, Kostić M, Milasin J. Estimation of total bacteria by real-time PCR in patients with periodontal disease. Srp Arh Celok Lek. Jan-Feb 2016;144(1-2):10-4. doi:10.2298/sarh1602010b
- 21. Mijailovic I, Nikolic N, Djinic A, et al. The down-regulation of Notch 1 signaling contributes to the severity of bone loss in aggressive periodontitis. J Periodontol. Apr 2020;91(4):554-561. doi:10.1002/jper.18-0755



# University of Belgrade SCHOOL OF DENTAL MEDICINE

Dr Subotića Str. No 8, phone: +381 11 2685-288 e-mail: <a href="mailto:stomfak@rcub.bg.ac.rs">stomfak@rcub.bg.ac.rs</a>



# ETHIC COMMITEE

Nº 36/6

On the ground of request of Assist. Prof. Iva Milinkovic, Ethic Committee of the School of Dental Medicine University of Belgrade, on the day of February 13<sup>th</sup> 2020, hereby signs the following

# **AGREEMENT**

We hereby agree with the methodology of research suggested by Assist. Prof. Iva Milinkovic within the following study

Adjunctive effect of local and systemic antimicrobials in non surgical treatment of periodontitis grade II and III

Translation of the seal: University of Belgrade School oh dental medicine 1948, Belgrade President of the Ethic Committee

Assoc Prof. dr Natasa Nikolic Jakoba

(signature)

Belgrade, March 10th 2020.